CLINICAL TRIAL: NCT03193229
Title: MapTrek, an Interactive, m-Health Intervention to Increase Activity Among Patients at Risk for Type 2 Diabetes
Brief Title: MapTrek to Increase Activity Among Patients at Risk for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Polgreen (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Philip Polgreen, Associate Professor of Medicine and Epidemiology; Director of Innovation Lab for Signal Center for Clinical Innovation, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201505733; 1R21DK108019-01A1 (NIH)
Record Dates: First submitted 2017-06-13; First posted 2017-06-20 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Pre Diabetes; Obesity
MeSH Terms: conditions — Glucose Intolerance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MapTrek (Experimental): Patients in the intervention group receive a Fitbit and MapTrek, an interactive text-messaging platform. The only equipment needed is a Fitbit (we provide) and a smartphone (required prior to enrollment). Each week, patients are assigned to a virtual walking route. Each day, they receive a text message with a link to the current route. The link will take them to a map where they can see their progress and the progress of others. A leaderboard provides information on how many steps each participant has taken. MapTrek also supports Street View on Google Maps, so patients can explore what they would see if they were in that location. Throughout each race, patients will randomly receive challenge text messages. Completing a challenge awards bonus steps to propel their character along the map.
  Interventions: Behavioral: MapTrek; Device: Fitbit
- Fitbit Only (Active Comparator): Patients randomized to the control group will receive a Fitbit only. This will allow us to determine if changes in physical activity are due to MapTrek or simply by giving the patients a Fitbit.
  Interventions: Device: Fitbit

INTERVENTIONS:
Behavioral: MapTrek — The objective of the study is to provide an inexpensive and scalable m-health tool to increase both volume and intensity of physical activity and reduce sedentary behavior in patients at risk for or already diagnosed with pre-diabetes.
  Arms: MapTrek
Device: Fitbit — Fitbit

SUMMARY:
The overarching objective of our work is to provide an inexpensive and scalable m-health tool to increase both volume and intensity of physical activity and reduce sedentary behavior in patients at risk for type 2 diabetes. The objective of this study is to pilot test MapTrek, a text-messaging based intervention.

DETAILED DESCRIPTION:
This study will randomize participants to 2 groups, an intervention group that will receive a Fitbit and MapTrek, and a control group that will receive a Fitbit only. This study has 3 specific aims.

Aim 1- To determine if patients randomized to MapTrek walk more than the control patients.

Aim 2- To determine if patients randomized to MapTrek generally walk at a faster pace during the day than control patients.

Aim 3- To determine if patients randomized to MapTrek have less sedentary time during the day than the control patients.

We expect to collect sufficient data to demonstrate the effectiveness of MapTrek, our prototype m-health tool, as an intervention to increase physical activity, heighten intensity of activity, and reduce sedentary behavior among a cohort of patients at risk for type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* English speaker
* Have a smart phone with texting and internet capabilities
* No aversion to research studies
* No active mental health conditions
* 1) Have a BMI > or equal to 25 and a history of hemoglobin A1C level between 5.7 and 6.4%, or 2) have a BMI > or equal to 30.

Exclusion Criteria:

* Pregnancy
* Prisoner status
* Taking insulin or other diabetic medications

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Total number of steps per day | 6 months
  The Fitbit will provide the total number of steps that each patient has taken per day.

SECONDARY OUTCOMES:
Pace of steps per day | 6 months
  The Fitbit will provide the number of steps taken per minute (pace) per day.

OTHER OUTCOMES:
Sedentary minutes per day | 6 months
  The Fitbit will provide the number of minutes spent being sedentary per day.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Polgreen, MD, Principal Investigator — Associate Professor of Infectious Diseases and Director of Signal Center for Clinical Innovation
Locations (1):
- Signal Center Innovation Lab, Coralville, Iowa, United States

IPD SHARING:
Plan to Share IPD: No